CLINICAL TRIAL: NCT02136381
Title: Pilot Randomised Controlled Trial of an Internet-based Lifestyle Intervention for People Around Retirement
Brief Title: Lifestyle Interventions at Retirement
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Newcastle University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: LiveWell_00745/2014
Record Dates: First submitted 2014-04-28; First posted 2014-05-13 (Estimated); Last update posted 2014-05-13 (Estimated); Status verified 2014-05

CONDITIONS: Health Behavior
Keywords: Lifestyle, interventions, retirement
MeSH Terms: conditions — Health Behavior

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- LEAP intervention (Experimental): A newly developed internet-based lifestyle programme (Living, Eating, Activity and Planning through retirement (LEAP)) will promote three key health and social behaviours; healthy eating following a Mediterranean diet, increasing physical activity and improve social connectedness.
  Interventions: Behavioral: LEAP intervention
- Control (Other): Thirty participants will be randomised to a minimal intervention comparator condition, where participants will be emailed a direct link to the National Health Service (NHS) choices 'LiveWell' website (http://www.nhs.uk/LiveWell/Pages/Livewellhub.aspx).
  This website contains general information on improving life style and health.
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: LEAP intervention — LEAP has 5 modules of tools and resources. LEAP is personalised based on information provided at different stages. The user determines the modules to complete (skipping or revisiting modules). Users can choose among 8 animated mentors (4 female; 4 male) to guide them through the intervention.
  Users will provide demographic data, health-related information, and current lifestyles in order to tailor the advice to be received.
  Advice will focus on adopting elements of a Mediterranean dietary pattern, increase physical activity, and improve social connectedness.
  Participants will receive 1) Mediterranean diet recipes; 2) a step counter to monitor physical activity goals; 3) advice in how to enhance social engagement and facilitate social roles
  Arms: LEAP intervention
Behavioral: Control — Thirty participants will be randomised to a minimal intervention comparator condition, where participants will be emailed a direct link to the National Health Service (NHS) choices 'LiveWell' website (http://www.nhs.uk/LiveWell/Pages/Livewellhub.aspx).
  The email will encourage the participants to access the health resources and information on the pages labelled men's health 40-60, men's health 60-plus, women's health 40-60, women's health 60-plus, as appropriate.
  Participants in the control group will be assessment after two months.
  Arms: Control

SUMMARY:
The LiveWell research programme aims to develop evidence-based, acceptable and scalable interventions to improve health and wellbeing in the retirement transition.

Life stage transitions involve changes in lifestyle and thus present key opportunities for behaviour change interventions. Our assessment of the literature shows that interventions with people of retirement age can effectively promote components of the Mediterranean diet (Lara et al, BMC Medicine Apr 8;12(1):60: 2014), physical activity (Hobbs et al, BMC Medicine Mar 19;11:75; 2013) and explicit social roles (Heaven et al, Milbank Q. Jun;91(2):222-87: 2013).

This study is a 2-month randomised controlled trial (RCT) with two intervention arms taking place in the North-East of England.

We have developed an internet-based lifestyle programme (Living, Eating, Activity and Planning through retirement (LEAP)) that promotes three key health and social behaviours; 1) healthy eating by adopting a Mediterranean diet, 2) increasing physical activity with the use of a step-counter, and 3) improving social connectedness.

Participants recruited for this study will be allocated in random order with a ratio of 2:1 to the intervention group (LEAP) or to a control group.

This study will evaluate the feasibility and acceptability of the LEAP intervention among people of retirement age and will pilot trial procedures.

In this programme of research we have also defined a suite of outcome measures and identified tools appropriate for capturing the Healthy Ageing Phenotype (HAP) (Lara et al, Maturitas. 2013 Oct;76(2):189-99). We will assess aspects of Cognition, Physical capability, Physiological outcomes, and psycho-social wellbeing. The feasibility and acceptability of these measures has yet to be determined and therefore will be formally assessed in this pilot RCT alongside more proximal outcomes of the intervention modules (i.e. diet, physical activity and social roles).

The hypotheses to be tested in the LiveWell programme are as follows:

* A newly developed internet-based lifestyle programme (Living, Eating, Activity and Planning through retirement (LEAP)) is an acceptable tool for behaviour change among people of peri-retirement age.
* A suite of outcome measures and identified tools appropriate for capturing the Healthy Ageing Phenotype (HAP) is acceptable among people of peri-retirement age.

DETAILED DESCRIPTION:
This intervention will last two months.

Participants will attend a 2-hour session with the researchers in order to provide signed consent and undergo the baseline assessment of healthy-ageing related outcome measures. Participants will attend a second 2-hour session after two months to repeat the assessment.

The assessments will take place at the participant's place of work. Participants who have retired will be asked to attend assessments at their previous place of work, at a local privately hired venue (e.g. community hall), or in their own homes.

Semi-structured interviews (n=28) will be conducted with a sample of participants from the intervention and control groups and two 'reduced participation' groups.

The reduced participation groups will include people who decline to participate in the trial but consent to a brief qualitative interview about their decision not to participate (after initially expressing interest) (n= up to 2), and people who withdraw from the trial but consent to a follow-up interview (n= up to 2).

The interviews will address three overlapping domains of enquiry: 1) questions relating to participation in the pilot study; 2) questions relating to use of the intervention website; and 3) questions relating to the use of the HAP set of measurement tools.

ELIGIBILITY:
Inclusion Criteria:

* Adults within 2 years (before/after) retirement from full time work
* Healthy volunteers
* Internet users
* English language speakers

Exclusion Criteria:

* Non-internet users
* Non-English speakers
* Not within the peri-retirement period (within two years of retirement)

Ages: 55 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2014-05; Primary Completion 2015-02 (Estimated); Study Completion 2015-02 (Estimated)

PRIMARY OUTCOMES:
Feasibility and acceptability of intervention | 2 months
  Participants will complete a questionnaire directed to obtain early markers of how the intervention is used

SECONDARY OUTCOMES:
Functional outcomes | At 0 and 2 months
  At baseline and at 2 months post-randomisation, participants will be asked to complete a series of tests to assess the impact of the programme on the following health-related indices:
  1. Resting blood pressure
  2. Lung function by spirometry (a breathing test measuring how much air someone can breathe in and out. It also measures how fast you can blow air out)
  3. Dexterity test (measuring the ability to coordinate fingers to manipulate objects quickly and accurately)
  4. Handgrip strength (a measure of muscle strength)
  5. Walking speed (measured by walking 4 meters at a normal pace)
  6. Endurance (measured by walking at a fast pace for 2 minutes)
  7. Standing balance
  8. Sit-to-stand test
  9. Timed-up-and-go test
  10. Cognitive function tests (such as memory and attention tests completed on a touchscreen computer)
  11. Psycho-social wellbeing tests (completed on a computer).
Change from baseline physical activity levels at 2 months | 0 and 2 months
  Physical activity will be assessed assessed during seven days at baseline and after 2 months interventions by accelerometry.
Change from baseline dietary intake | 0 and 2 months
  Participants will self-report dietary intake using the 24-hour dietary recall method. Three days (including 2 weekdays and 1 weekend day) of dietary intake at baseline and after two months will be reported.
Change from baseline resting blood pressure at 2 months | 0 and 2 months
Change from baseline lung function at 2 months | 0 and 2 months
  Lung function will be measured by spirometry (a breathing test measuring how much air someone can breathe in and out. It also measures how fast you can blow air out)
Change from baseline dexterity at 2 months | 0 and 2 months
  The National Institutes of Health Toolbox dexterity test, involving the 9-hole pegboard test (measuring the ability to coordinate fingers to manipulate objects quickly and accurately), will be used.
Change from baseline Handgrip strength at 2 months | 0 and 2 months
Change from baseline walking speed at 2 months | 0 and 2 months
  Walking speed will be measured by walking 4 meters at a normal pace
Change from baseline endurance at 2 months | 0 and 2 months
  Endurance will be measured as the total distance walked at a fast pace during 2 minutes
Change from baseline standing balance at 2 months | 0 and 2 months
Change from baseline functional change of transitional movements at 2 months | 0 and 2 months
  The sit-to-stand test will be used
Change from baseline mobility at 2 months | 0 and 2 months
  The timed-up-and-go test will be used
Change from baseline episodic memory at 2 months | 0 and 2 months
  The Paired Associates Learning (PAL) episodic memory test will be used
Change from baseline verbal and category fluency at 2 months | 0 and 2 months
  The verbal and category fluency test will be used
Change from baseline processing speed at 2 months | 0 and 2 months
  The letter digit substitution test will be used
Change from baseline life satisfaction at 2 months | 0 and 2 months
  The satisfaction with life scale will be used
Change from baseline quality of life at 2 months | 0 and 2 months
  The World Health Organization Quality of Life scale (WHOQoL-BREF) will be used
Change from baseline meaning and purpose at 2 months | 0 and 2 months
  The National Institutes of health toolbox meaning and purpose test will be used
Change from baseline social companionship at 2 months | 0 and 2 months
  The companionship scale of the Patient-Reported Outcomes Measurement Information System (PROMIS) will be used
Change from baseline emotional support at 2 months | 0 and 2 months
  The Patient-Reported Outcomes Measurement Information System (PROMIS) emotional support scale will be used
Change from baseline social functioning at 2 months | 0 and 2 months
  The Patient-Reported Outcomes Measurement Information System (PROMIS) Satisfaction with social roles scale will be used
Acceptability, feasibility and compliance with the healthy ageing phenotype (HAP) battery assessment procedures | 2 months
  Participants will complete a questionnaire directed to evaluate the acceptability, feasibility and compliance with the healthy ageing phenotype (HAP) battery assessment procedures
Change from baseline positive affect at 2 months | 0 and 2 months
  The National Institutes of Health toolbox "positive affect scale" will be used
Change from baseline instrumental support at 2 months | 0 and 2 months
  The National Institutes of Health toolbox "instrumental support" scale will be used
Change from baseline satisfaction with social roles and activities at 2 months | 0 and 2 months
  The National Institutes of Health toolbox "satisfaction with social roles and activities" scale will be used.
Change from baseline social isolation at 2 months | 0 and 2 months
  The National Institutes of Health toolbox "social isolation" scale will be used
Change from baseline depression scale at 2 months | 0 and 2 months
  The Center for Epidemiologic Studies Depression Scale (CES-D) will be used

CONTACTS AND LOCATIONS:
Overall Officials: John C Mathers, PhD, Study Director — Human Nutrition Research Centre, Institute for Ageing and Health, Newcastle University; Martin White, PhD, Principal Investigator — Institute for Health and Society, Newcastle University; Falko F Sniehotta, PhD, Principal Investigator — Institute for Health and Society, Newcastle University; Lynn Rochester, PhD, Principal Investigator — Newcastle University; Moynihan J Paula, PhD, Principal Investigator — Newcastle University; Thomas D Meyer, PhD, Principal Investigator — Institute of Neuroscience, Newcastle University
Locations (1):
- Human Nutrition Research Centre, Institute for Ageing and Health, Newcastle University, Newcastle upon Tyne, Tyne and Wear, United Kingdom

REFERENCES:
- [Derived] Lara J, O'Brien N, Godfrey A, Heaven B, Evans EH, Lloyd S, Moffatt S, Moynihan PJ, Meyer TD, Rochester L, Sniehotta FF, White M, Mathers JC. Pilot Randomised Controlled Trial of a Web-Based Intervention to Promote Healthy Eating, Physical Activity and Meaningful Social Connections Compared with Usual Care Control in People of Retirement Age Recruited from Workplaces. PLoS One. 2016 Jul 29;11(7):e0159703. doi: 10.1371/journal.pone.0159703. eCollection 2016. PMID 27472560